## Ultraslow full-power SWL versus slow power-ramping SWL in stones with high attenuation value

Document Date: September 1, 2015

## Statistical analysis:

- SPSS version 15
- Intention-to-treat approach
- The two groups compared in all perioperative data including the criteria of patients and stones, number of sessions and SW, success rate and the complications using Student-t test for normally distributed continuous variables or Mann-Whitney test for non parametric data. Categorical variables were analysed using Chi-square test or Fisher-Exact test.
- A two sided p < 0.05 was considered significant.
- Sample size calculation was performed for the primary outcome (stone clearance).